CLINICAL TRIAL: NCT06523374
Title: Endoscopic Brush Cytology and Single Cell Clonal Dynamics of Early Esophageal Adenocarcinoma for Defining Cost Effective Surveillance Strategies and Prediction of Cancer Recurrence: Prospective Pilot Cohort Study in Preparation of a Randomized Controlled Trial to Determine the Feasibility of a Risk Stratification Model for Barrett Esophagus Patients Based on Brush Cytology, and to Test Novel High Throughput Methods for Assessing Biomarkers for Future Use
Brief Title: A Study of Barrett's Esophagus Patients to Investigate Quality of Life and Fear of Cancer, and Optimize a Risk Model Based on Biomarkers and New Technologies to Better Predict the Development of Cancer
Acronym: Endeavor-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Karolinska Institutet (Other); Universal Diagnostics (Industry); Amsterdam UMC (Other); Radboud University Medical Center (Other); AZ Delta (Other); Centre Hospitalier Universitaire de Liege (Other); University of Leipzig (Other); IRCCS Ospedale San Raffaele (Other); Karolinska University Hospital (Other); University of Dublin, Trinity College (Other); Heinrich-Heine University, Duesseldorf (Other); GZA Ziekenhuizen Campus Sint-Augustinus (Other); University Hospital, Ghent (Other); Rigshospitalet, Denmark (Other); Universitätsklinikum Leipzig (Other); St. James's Hospital, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDGE3788; 101136935 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2024-06-17; First posted 2024-07-26 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Barrett's Esophagus; Esophageal Adenocarcinoma
Keywords: Barrett; Barrett's Esophagus; Endeavor; Esophageal cancer; Esophageal adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic brush cytology (Other): Each participant will receive all interventions. A routine endoscopy will be planned during which several minimally invasive interventions will be performed:
  drawing a blood sample (standard of care), brush cytology (not standard of care) and biopsies (standard of care) during the endoscopy.
  Interventions: Procedure: Endoscopic brush cytology

INTERVENTIONS:
Procedure: Endoscopic brush cytology — A total of four brush samples will be taken during the endoscopy. Other minimally invasive interventions during this study are standard of care.

SUMMARY:
This study serves, in part, to prepare for a future large cohort study. The goal of the study is:

1. The collection of various tissue samples (blood, biopsies and "esophageal brushes") and their analysis.
2. To set up standardized methods for different genetic analyses (DNA-FISH and so-called single cell sequencing) on the esophageal tissue samples.
3. Evaluating the quality of life of Barrett's Esophagus patients and the degree of fear of getting cancer.

Patients with a Barrett's Esophagus can participate in the study if they are minimally 18 years old, are capable of giving informed consent (fully understanding what the study entails before giving consent to participate), have Barrett Esophagus and are referred to one of the participating centers due to suspicion of high-grade dysplasia or early esophageal cancer, for which the participant will be evaluated by endoscopic imaging and biopsy.

Study procedures:

* An intake consultation will be planned, wherein the eligibility criteria will be assessed, and participant characteristics will be collected.
* A routine gastroscopy will be planned twice during which several minimally-invasive interventions will be performed: drawing a blood sample, brush cytology during the endoscopy (a brush is used to obtain cells from the surface of the esophagus) and obtaining biopsy samples (small pieces of tissue). Each participant will need to undergo all the interventions.
* Patients will have to complete questionnaires at three time points to assess their quality of life (EQ-5D-DL questionnaire) and fear of cancer recurrence (Cancer Worry Scale).

DETAILED DESCRIPTION:
More specifically, you will have a standard endoscopy twice during which tissue samples will be taken from the esophagus to check for the severity of the disease. This is part of standard care. If you participate in the study, additional samples will be taken from the esophagus and also from the stomach (a total maximum of 10 samples of 1-2 mm). As a result, the endoscopic examination will take about 10-15 minutes longer than standard. Furthermore, in addition to the tissue samples, cells of the esophageal mucosa will be sampled (through 4 "esophageal brushes") and blood (4 tubes) will also be collected.

For this study, you will be contacted a total of three times. Once for a screening visit and twice for the sample collection described above. The screening and sample collection will take place during the already scheduled treatments and consultations. Afterwards, patient outcomes will be documented for the study until a maximum of 5 years after inclusion. This documentation will take place during the routine follow up so does not require any additional visits for the patients. Additionally you will be asked to complete two short questionnaires on your mobile phone at three time points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known BE undergoing endoscopy for possible treatment by EMR or ESD due to suspicion of early esophageal Barrett cancer
* Capable of receiving informed consent and of giving permission
* Age 18 and upward

Exclusion Criteria:

* Patients with current known malignancy of the gastrointestinal tract other than the esophageal lesion
* Patients with severe co-morbidity that prohibits endoscopic therapy under sedation or conscious sedation (such as severe cardiac or pulmonary disease)
* Esophageal varices
* Uncontrollable coagulation disorders
* Undergoing chemotherapy or immunotherapy or received chemotherapy < 6 weeks prior to endoscopy
* Undergoing radiotherapy within the esophageal region or received chemotherapy < 6 months prior to endoscopy
* WHO score > 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of brush, biopsy and blood samples obtained from different sites for analysis by HTP technologies | 6-12 months
  We will determine the success rate of obtaining material from different sites for analysis by high throughput technologies (Next Generation Sequencing) of the brush, biopsy or blood samples. A rate of analysable cells of at least 80% of the specimens will be regarded as successful.
Success rate of DNA-FISH analyses on the brush cytology samples | 6-12 months
  Our second primary outcome measure for this pilot study is successful DNA-FISH analysis (successful = at least 50 cells that can be analyzed in at least 80% of participants) on the brush cytology samples for defining the final risk model that will be applied in the randomized controlled trial following the pilot study.

SECONDARY OUTCOMES:
Accuracy of a DNA-FISH based risk model | 6-24 months
  The first secondary outcome is the accuracy of a DNA-FISH based risk model to distinguish low risk from high-risk early Barrett cancers. This will be assessed by endoscopic imaging and histo-pathological outcomes.
Correlation of a DNA-FISH based risk model | 6-24 months
  The correlation of a DNA-FISH based risk model to distinguish low risk from high-risk early Barrett cancers with results obtained from Next Generation Sequencing.
Standard operating procedures for specimen collection | 6-24 months
  A standard operating procedure describing the best method for obtaining brush cytology specimens and for obtaining the right tissue specimens via endoscopy will be created. The best method will be determined by the quality and number of analysable cells.
Standard operating procedures for logistical procedures | 6-24 months
  A standard operating procedure (SOP) for the logistics for shipment, redistribution and storage of patient material and data of the different participating sites will be created based on the course of this pilot study. Interim logistical problems will be spontaneously reported by all sites and resolved with the central team. The final solutions ("best method") will be described in the SOP.
Successful participation and answering of questionnaires | 6-24 months
  The participation and answering of the quality of life questionnaires and anxiety level questionnaires of at least 70% of the patients will be seen as successful.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Krishnadath, Principal Investigator — Universitair Ziekenhuis Antwerpen (UZA)
Locations (9):
- Belgium (4):
  - University Hospital Antwerp, Edegem, Antwerpen
  - Sint-Augustinus Hospital (ZAS), Wilrijk, Antwerpen
  - UZ Gent, Ghent
  - AZ Delta, Roeselare
- Rigshospitalet, Copenhagen, Denmark
- CHU LILLE - Centre Hospitalier Universitaire de Lille, Lille, France
- St James's Hospital, Dublin, Ireland
- IRCCS Ospedale San Raffaele, Milan, Milano, Italy
- Karolinska University Hospital, Solna, Sweden